CLINICAL TRIAL: NCT03560453
Title: Facilitating Employment for Youth With Autism: A Replication Study of an Internship Model to Identify Evidence Based Practices
Brief Title: Facilitating Employment for Youth With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM15031; NIDILRRDRRP13-16 (Other Grant/Funding Number: Natnl. Inst. Disability Independent Living Rehabilitation Research)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Autism Spectrum Disorder; Autism; Asperger Syndrome; Pervasive Developmental Disorder; Adolescent Development
Keywords: Autism; ASD; Competitive Integrated Employment; Project SEARCH; Outcomes; Support Intensity
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive

STUDY DESIGN:
Intervention Model Description: Non-pharmacologic randomized clinical trial and followed the Non-pharmacological Consolidated Standards of Reporting Trials Statement recommendations to conduct the research (CONSORT; Boutron, Altman, Moher, Schulz, & Ravaud, 2017)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Attend assigned high school for 9 months
- Project SEARCH plus ASD Supports (Experimental): Attend Project SEARCH plus ASD Supports for 9 months
  Interventions: Behavioral: Project SEARCH Plus ASD Supports

INTERVENTIONS:
Behavioral: Project SEARCH Plus ASD Supports — Project SEARCH is an intensive 9-month job training program where youth with developmental disabilities in their last year of high school are embedded in a large community business such as a hospital, government complex, or banking center (Daston et al., 2012). Students with developmental disabilities who participate in this model rotate through three 10-12 week internships within the business where they log approximately 720 hours of internship time learning marketable skills while receiving supported employment. They also get 180 hours of classroom time at the business for a total of approximately 900 hours embedded in the business setting. In addition to these important training components, Project SEARCH requires collaboration between multiple community partners to support students in attaining employment upon completion of the program. Collaborations include students with developmental disabilities and their family, a LEA, a local CRP, the state VR, and a host business.
  Other Names: PS+ASD
  Arms: Project SEARCH plus ASD Supports

SUMMARY:
This study will test the efficacy of a nationally recognized employment training and placement program (Project SEARCH) when applied to youth with Autism Spectrum Disorders. It is designed to examine a single overall research question:

Research Question: To what extent does a collaborative, employer-based employment training and placement program improve the employment outcomes, need for support, social responsiveness, self-determination, and quality of life of young adults with ASD 18-21 served in public special education programs?

DETAILED DESCRIPTION:
In this project, the investigators propose testing the efficacy of the Project SEARCH model that has been successfully implemented for youth with ASD at one site in a 300-bed hospital in Richmond, VA. The investigators will accomplish this by continuing the Project SEARCH study that has been implemented for youth with ASD and expanding this model to two additional sites in Virginia. The investigators also propose expanding the current randomized clinical trial protocol to the two new sites. In doing so, the investigators will be able to further develop the model while also assessing the strength of the relationship between the intervention and outcomes achieved. Additionally, the investigators will identify programmatic and individual factors that affect successful employment outcomes as well as other critical behaviors that are essential for youth with ASD to exhibit such as socialization, communication, independence and self management. Finally, through the proposed project the investigators will be able to provide evidence to guide decisions related to fidelity of implementation of the components necessary to replicate Project SEARCH for youth with ASD.

Hypotheses: There are one primary and six secondary endpoints under investigation in the proposed study: (1) Employment status upon completion of the program, 90 days post completion, and 12 months post completion (primary); (2) wage upon completion, 90 days post completion, and 12 months post completion; and (3) number of hours worked per week upon completion, 90 days post completion, and 12 months post completion. In addition, the effect of the intervention on (4) student support needs, (5) social responsiveness, and (6) self-determination will be explored. Hypotheses related to these endpoints, or dependent variables, include:

* Hypothesis I -- Young adults who participate in an employer-based employment training and placement program will demonstrate a higher rate of employment than those in the control condition.
* Hypothesis II -- Young adults who participate in a work-based employment training and placement program will earn higher wages on average at project completion compared to those in the control condition.
* Hypothesis III -- Young adults who participate in a work-based employment training and placement program will work more hours per week on average than those in the control condition.
* Hypothesis IV -- Young adults who participate in a work-based employment training and placement program will reduce their need for employment supports compared to those in the control condition, as measured by the Employment Subscale of the Support Intensity Scale.
* Hypothesis V -- Young adults who participate in a work-based employment training and placement program will increase their social responsiveness skills compared to those in the control condition, as measured by the Social Responsive Scale (SRS-2).
* Hypothesis VI -- Young adults who participate in a work based employment training and placement program will increase their self-determination skills compared to those in the control condition, as measured by the Arc's Self-Determination Scale (Adolescent Version).
* Hypothesis VII - Young adults who participate in a work based employment training and placement program will increase their quality of life compared to those in the control condition, as measured by the Quality Metrics Health Outcomes SF-36v2.

ELIGIBILITY:
Inclusion Criteria: (1) student in a local public school where the research was being conducted, (2) had a medical diagnosis of ASD or educational identification of autism, (3) was between the ages of 18-21 on the first day of the next school year, (4) displayed independent self-care, including using the bathroom, eating, and moving from place to place independently (5) had eligibility for funding through the state vocational rehabilitation agency, and (6) had continued eligibility for public school services -

Exclusion Criteria: Unable to provide consent or assent

-

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Employment Outcomes Survey from Graduation to 12 months follow-up | Graduation and 12 month follow-up
  Employment status (Employed Full-Time, Employed Part-Time, Not Employed/Looking for Employment, and Not Employed/Not Looking for Employment) will be measured at the point of graduation and 12 months follow-up. At these data collection points we will also collect information on hourly wage, changes in hourly wage, hours worked per week (or per month if the individual works a variable schedule), and fringe benefits received, including annual or sick leave, medical/dental benefits, retirement benefits, life insurance, and health and wellness. This is a researcher developed survey

SECONDARY OUTCOMES:
Change in the Support Intensity Scale (SIS; Thompson, et al., 2004) from Graduation to 12 months follow-up | Baseline, Graduation and 12 month follow-up
  The Supports Intensity Scale (SIS, Thompson, et al., 2004) is an interview based assessment tool that identifies the type, amount, and frequency of support required by individuals with significant disabilities, including persons with autism, to perform 57 life activities. An additional 28 items address behavioral and medical areas. The assessment is completed through an interview with the individual, as well as family, school, and community members with in-depth knowledge of the individual. The assessment generates a composite scale score and individual scale scores in the areas of home living, community living, lifelong learning, employment, health and safety, and social areas. The Composite Scale Score and the Employment Subscale Score will be used as dependent measures. Scores are presented as t-scores and are compared to a normed population of individuals with disabilities.
Change in Social Responsiveness Scale, Second Edition (Constantino & Gruber, 2012) from Graduation to 12 months follow-up | Baseline, Graduation, and 12 month follow-up
  The Social Responsiveness Scale, Second Edition (SRS-2), (Constantino & Gruber, 2012) will be used to measure the effect of the treatment intervention in comparison to the control condition on subject's social awareness, social cognition, social communication and social motivation. It will be used at all four points of data collection to measure changes that occur in the individual's ability in social interactions and verbal discussions in social situations. The SRS-2 is a 65-item scale that has been used as a measure of treatment effectiveness in recent studies (Booker & Starling, 2011; Aldridge, Gibbs, Schmidhofer, & Williams, 2012; Gantman, Knapp, Orenski & Laugeson, 2012). Scores are presented as t-scores and are compared to a normed population of individuals with ASD.
Change in The ARC's Self-Determination Scale (Wehmeyer, 1996) from from Graduation to 12 months follow-up | Baseline, Graduation, and 12 month follow-up
  The Arc's Self-Determination Scale (Wehmeyer, 1996b; Wehmeyer & Kelchner, 1995) is a 72-item self-report scale that provides data on overall self-determination by measuring individual performance in the four essential characteristics of self-determined actions including autonomy, self-regulation, psychological empowerment, and self-realization. These four characteristics are subscales within the Scale. The Scale generates a total Self-Determination score as well as scores for the four subtests. The total score on the Scale will serve as a dependent measure for the proposed study. Scores are presented as t-scores and are compared to a normed population of people with and without disabilities.
Change in The Short Form 36 Version 2 (SF-36v2, Maurish & Turner-Bowker, 2009) from from Graduation to 12 months follow-up | Baseline, Graduation, and 12 month follow-up
  The SF-36v2 Health Survey is a 36 item questionnaire used to measure eight domains of health-related quality of life including Physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health. The information obtained from these eight health domains are further aggregated into two summary measured: the physical component summary, and the mental component summary. Data from the survey will be used to compare health outcomes between the two groups health status. It will be used in this study to measure health outcomes between the treatment and control group. Scores are presented as t-scores and are compared to a normed population of people without disabilities.

CONTACTS AND LOCATIONS:
Overall Officials: Carol M Schall, PhD, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wehman P, Schall C, Carr S, Targett P, West M, Cifu G. Transition from school to adulthood for youth with ASD: what we know and what we need to know. J Disabil Policy Stud. 2014;25:30-40. doi:10.1177/1044207313518071.
- [Result] Schall C, Wehman P, McDonough JL. Transition from school to work for students with autism spectrum disorders: understanding the process and achieving better outcomes. Pediatr Clin North Am. 2012 Feb;59(1):189-202, xii. doi: 10.1016/j.pcl.2011.10.009. PMID 22284802
- [Result] Wehman PH, Schall CM, McDonough J, Kregel J, Brooke V, Molinelli A, Ham W, Graham CW, Erin Riehle J, Collins HT, Thiss W. Competitive employment for youth with autism spectrum disorders: early results from a randomized clinical trial. J Autism Dev Disord. 2014 Mar;44(3):487-500. doi: 10.1007/s10803-013-1892-x. PMID 23893098
- [Result] Schall CM, Wehman P, Brooke V, Graham C, McDonough J, Brooke A, Ham W, Rounds R, Lau S, Allen J. Employment Interventions for Individuals with ASD: The Relative Efficacy of Supported Employment With or Without Prior Project SEARCH Training. J Autism Dev Disord. 2015 Dec;45(12):3990-4001. doi: 10.1007/s10803-015-2426-5. PMID 25791125
- [Result] Wehman P, Schall CM, McDonough J, Graham C, Brooke V, Riehle JE, Brooke A, Ham W, Lau S, Allen J, Avellone L. Effects of an employer-based intervention on employment outcomes for youth with significant support needs due to autism. Autism. 2017 Apr;21(3):276-290. doi: 10.1177/1362361316635826. Epub 2016 Jul 9. PMID 27154907
- [Derived] Schall C, Sima AP, Avellone L, Wehman P, McDonough J, Brown A. The Effect of Business Internships Model and Employment on Enhancing the Independence of Young Adults With Significant Impact From Autism. Intellect Dev Disabil. 2020 Aug 1;58(4):301-313. doi: 10.1352/1934-9556-58.4.301. PMID 32750714
- [Derived] Wehman P, Schall C, McDonough J, Sima A, Brooke A, Ham W, Whittenburg H, Brooke V, Avellone L, Riehle E. Competitive Employment for Transition-Aged Youth with Significant Impact from Autism: A Multi-site Randomized Clinical Trial. J Autism Dev Disord. 2020 Jun;50(6):1882-1897. doi: 10.1007/s10803-019-03940-2. PMID 30825082
- See also: This website provides a link to numerous research briefs, webinars, and webcasts developed to describe the project — http://vcurrtc.org/school2work/

DOCUMENTS (4):
  • Informed Consent Form: Student Consent Form (2015-04-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT03560453/ICF_000.pdf
  • Informed Consent Form: Student Assent Form (2015-04-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT03560453/ICF_001.pdf
  • Informed Consent Form: Educator Consent (2015-04-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT03560453/ICF_002.pdf
  • Informed Consent Form: LAR Consent (2015-04-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT03560453/ICF_003.pdf